CLINICAL TRIAL: NCT02232243
Title: A Pilot Study to Determine the Biological Effects of Hydroxychloroquine on PAR-4 Levels in Patients With Resectable Solid Tumors
Brief Title: HCQ on PAR-4 Levels in Patients With Resectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peng Wang, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Peng Wang, MD PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-MULTI-14-MCC
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor
Keywords: Cancer; Surgery; Hydroxychloroquine
MeSH Terms: conditions — Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Initial: Hydroxychloroquine 400mg HCQ (Experimental): These initial 3 patients received 200mg hydroxychloroquine (HCQ) twice daily (400mg/day total) for 14 days prior to surgery.
  Interventions: Drug: Hydroxychloroquine, 200mg twice dailiy
- Secondary: Hydroxychloroquine 800mg HCQ (Experimental): Based on data analysis from the initial patients, these patients received 400mg hydroxychloroquine (HCQ) twice daily (800mg/day total) for 14 days prior to surgery.
  Interventions: Drug: Hydroxychloroquine, 400mg twice daily
- Tertiary: Hydroxychloroquine 400mg HCQ (Experimental): Based on data from the primary and secondary groups, patients received 200mg hydroxychloroquine (HCQ) twice daily (400mg/day total) for 14 days prior to surgery.
  Interventions: Drug: Hydroxychloroquine, 200mg twice dailiy

INTERVENTIONS:
Drug: Hydroxychloroquine, 200mg twice dailiy — Hydroxychloroquine, 200mg twice daily (400mg/day total) was given to subjects for up to 14 days prior to surgery.
  Arms: Initial: Hydroxychloroquine 400mg HCQ; Tertiary: Hydroxychloroquine 400mg HCQ
Drug: Hydroxychloroquine, 400mg twice daily — Hydroxychloroquine, 400mg twice daily (800mg/day total) was given to subjects for up to 14 days prior to surgery.
  Arms: Secondary: Hydroxychloroquine 800mg HCQ

SUMMARY:
Baseline levels of PAR-4 secreted by normal cells are generally inadequate to cause massive apoptosis in cancer cells and drugs that bolster the secretion of PAR-4 would constitute an important therapeutic advance.The apoptosis sensitizing features of hydroxychloroquine enhance the anti-tumor effects of a broad range of cancer therapeutics. The investigators hypothesize that hydroxychloroquine will induce at least 2-fold increase in systemic (plasma) PAR-4 levels compared to pre-treatment plasma levels in patients with resectable solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed solid tumor that is planned for surgical resection.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must be able to ingest oral medications.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin Less than 1.5 x ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Creatinine within normal institutional limits OR Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Patients must be able to undergo surgical resection of their tumor as determined by the treating surgeon.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with metastatic cancer and/or cancer that is not amenable to surgery.
* Patients with significant malabsorption as determined by the treating physician.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with primary brain tumors amenable to surgery are allowed on this protocol.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to hydroxychloroquine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with hydroxychloroquine. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients that are on enzyme-inducing anti-epileptic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, PhD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang P, Burikhanov R, Jayswal R, Weiss HL, Arnold SM, Villano JL, Rangnekar VM. Neoadjuvant administration of hydroxychloroquine in a phase 1 clinical trial induced plasma Par-4 levels and apoptosis in diverse tumors. Genes Cancer. 2018 May;9(5-6):190-197. doi: 10.18632/genesandcancer.181. PMID 30603055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated July 2015 at the University of Kentucky and enrolled 10 adult patients with early stage solid malignancies.
Pre-assignment Details: 10 patients enrolled in this dose escalation study. In Period 1, three patients were assigned to receive 200mg HCQ twice daily. Based on toxicity and PAR-4 levels, in Period 2 the next four patients received 400mg HCQ twice daily. Following additional analysis, in Period 3 the final three patients received 200mg HCQ twice daily.
Groups:
- Initial: Hydroxychloroquine 400mg HCQ: These patients received 200mg hydroxychloroquine (HCQ) twice daily (400mg/day total) for 14 days prior to surgery.
- Secondary: Hydroxychloroquine 800mg HCQ: These patients received 400mg hydroxychloroquine (HCQ) twice daily (800mg/day total) for 14 days prior to surgery.
- Tertiary: Hydroxychloroquine 400mg HCQ: Based on data from primary and secondary groups, these patients received 200mg hydroxychloroquine (HCQ) twice daily (400mg/day total) for 14 days prior to surgery.
Period: First Dose (200mg HCQ Twice Daily)
Arm/Group | Initial: Hydroxychloroquine 400mg HCQ | Secondary: Hydroxychloroquine 800mg HCQ | Tertiary: Hydroxychloroquine 400mg HCQ
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Second Dose (400mg HCQ Twice Daily)
Arm/Group | Initial: Hydroxychloroquine 400mg HCQ | Secondary: Hydroxychloroquine 800mg HCQ | Tertiary: Hydroxychloroquine 400mg HCQ
Started | 0 | 4 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Period: Third Dose(200mg HCQ Twice Daily)
Arm/Group | Initial: Hydroxychloroquine 400mg HCQ | Secondary: Hydroxychloroquine 800mg HCQ | Tertiary: Hydroxychloroquine 400mg HCQ
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Initial: Hydroxychloroquine 400mg HCQ; Tertiary: Hydroxychloroquine 400mg HCQ: Hydroxychloroquine 14 days
  Hydroxychloroquine: Hydroxychloroquine (200mg twice per day; 400mg total) was given to subjects for up to 14 days prior to surgery.
- Secondary: Hydroxychloroquine 800mg HCQ: Hydroxychloroquine 14 days
  Hydroxychloroquine: Hydroxychloroquine (400mg twice per day; 800mg total) was given to subjects for up to 14 days prior to surgery.
- Total: Total of all reporting groups
Arm/Group | Initial: Hydroxychloroquine 400mg HCQ | Secondary: Hydroxychloroquine 800mg HCQ | Tertiary: Hydroxychloroquine 400mg HCQ | Total
Number analyzed (Participants) | 3 | 4 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: One patient was unanalyzable
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 2 | 3 | 3 | 8
    >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient was unanalyzable
  Participants
    Female | 0 | 0 | 1 | 1
    Male | 3 | 4 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One patient was unanalyzable
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 3 | 4 | 3 | 10
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: one patient unanalyzable
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 3 | 4 | 3 | 10
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Patients With Elevated Par-4 Levels
Description: Number of patients with 2-fold change in Par-4 levels from baseline to day 14
Time Frame: Baseline and day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Initial: Hydroxychloroquine 400mg HCQ | Secondary: Hydroxychloroquine 800mg HCQ | Tertiary: Hydroxychloroquine 400mg HCQ
Number analyzed (Participants) | 3 | 3 | 3
Participants | 3 | 2 | 1

2. Primary Outcome: Optimal Biologic Dose of Hydroxychloroquine
Description: Dose (mg twice daily) wherein 70% of patients exhibit a 2-fold increase in Par-4 levels with a dose-limiting toxicity of no more than 30%.
Time Frame: Day 14
Population: All patients
Measure: Number; unit: mg twice daily
Groups:
- All Patients: Optimal biological dose is calculated from aggregate data of all patients
Arm/Group | All Patients
Number analyzed (Participants) | 9
mg twice daily | 200

ADVERSE EVENTS:
Time Frame: 14 days
Description: Patients were queried about adverse events during study visits.
Groups:
- Initial: Hydroxychloroquine 400mg HCQ: Hydroxychloroquine 14 days
  Hydroxychloroquine: Hydroxychloroquine (200mg twice daily; 400mg total) was given to subjects for up to 14 days prior to surgery.
- Secondary: Hydroxychloroquine 800mg HCQ: Hydroxychloroquine 14 days
  Hydroxychloroquine: Hydroxychloroquine (400mg twice daily; 800mg total) was given to subjects for up to 14 days prior to surgery.
- Tertiary: Hydroxychloroquine 400mg HCQ: Hydroxychloroquine 14 days
  Hydroxychloroquine: Hydroxychloroquine (200mg twice daily, 400mg total) was given to subjects for up to 14 days prior to surgery.
Arm/Group | Initial: Hydroxychloroquine 400mg HCQ | Secondary: Hydroxychloroquine 800mg HCQ | Tertiary: Hydroxychloroquine 400mg HCQ
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 2/4 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial: Hydroxychloroquine 400mg HCQ (N=3) | Secondary: Hydroxychloroquine 800mg HCQ (N=4) | Tertiary: Hydroxychloroquine 400mg HCQ (N=3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT02232243/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT02232243/ICF_001.pdf